CLINICAL TRIAL: NCT00979342
Title: Interlace Medical Comparative Sedation Study
Brief Title: Comparative Sedation Study of the MyoSure Hysteroscopic Tissue Removal System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hologic, Inc. (Industry)
Responsible Party: John Vozella, V.P Clinical & Regulatory Affairs, Interlace Medical, Inc,
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMP 200902
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-07

CONDITIONS: Uterine Fibroids; Polyps
Keywords: morcellator; hysteroscope; myomectomy; polypectomy; uterine fibroids; uterine polyps; local anesthetic; cervical block; pain management
MeSH Terms: conditions — Leiomyoma; Polyps; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cervical Block, 6 injection sites (Experimental): Subject will receive a cervical block of 1% lidocaine and 0.25% bupivacaine, with injections in the following locations: 2cc at 12:00, 10cc at 3:00, 10 cc at 9:00, 5 cc at 4:00, 5 cc at 8:00, and 5 cc at 6:00.
  Interventions: Device: Hysteroscopic Morcellator
- Cervical Block, 2 injection sites (Experimental): Subject will receive a cervical block of 1% lidocaine and 0.25% bupivacaine, with injections in the following locations: 10 cc at 4:00, and 10 cc at 8:00.
  Interventions: Device: Hysteroscopic Morcellator
- Ibuprofen q. 8 hours (Experimental): Subjects will receive a post procedure pain management regimen of ibuprofen 800 mg every 8 hours, for the first 24 hours and then PRN.
  Interventions: Device: Hysteroscopic Morcellator
- Ibuprofen PRN (Experimental): Subjects will receive a post procedure pain management regimen of ibuprofen 800 mg PRN.
  Interventions: Device: Hysteroscopic Morcellator

INTERVENTIONS:
Device: Hysteroscopic Morcellator — The MyoSure Tissue Removal Device consists of a hand-held tissue removal device comprising a mechanical drive assembly connected to a drive cable and associated control box on one end, and a 3 mm shaft on the other end of the device. The shaft is approximately 12 cm long and equipped with an open channel that houses an oscillating blade.When the side channel is exposed to target tissue and the motor is activated, the oscillating blade will cut the tissue within the channel. Once cut, the tissue travels down the center of the 3mm shaft via suction coupled to the proximal end of the tissue removal device, and is trapped in a vacutainer bottle.
  Other Names: MyoSure Hysteroscopic Tissue Removal System; MyoSure Tissue Removal Device

SUMMARY:
The purpose of this study is to develop a recommended local anesthetic protocol and post-treatment pain management regimen, in order to assure patient comfort during office-based treatment with the MyoSure Hysteroscopic Tissue Removal Device. Subject self-reported pain scores (as rated on an 11 point scale) will be compared at multiple time intervals between all treatment groups.

DETAILED DESCRIPTION:
Forty subjects will be enrolled in a randomized, controlled study conducted at four physician offices or day surgery settings. Subjects will be randomized 1:1 to a local anesthetic group (Group #1 or Group #2). Subjects will undergo a hysteroscopic tissue removal procedure to remove intrauterine polyps, type 0 fibroids, or type I fibroids. Subsequent to the procedure, subjects will be randomized 1:1 within the local anesthetic group to a post procedure pain management group (Group A or Group B). Subject self-reported pain scores (as rated on an 11 point scale)will be compared at three time points: Immediately post procedure, prior to discharge from the treatment facility, and at 48 hours post procedure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female between the ages of 18 and 65
* Subject must be able to understand, read and sign the study specific informed consent forms after the nature of the study has been fully explained to her
* Subject is a pre-menopausal or peri-menopausal female, either nulliparous or parous
* Subject is indicated for myomectomy or polypectomy for benign pathology, based on hysteroscopic, ultrasound, or saline infused sonogram assessment within 60 days
* Subject exhibits intrauterine polyps and/or submucous myomas which meet one of the following criteria. In cases of subjects with multiple intrauterine pathology, classification is based as follows:

  * All polyps
  * A single Type 0 or Type 1 myoma ≤ 3 cm
  * Polyps plus a single Type 0 or Type 1 myoma ≤ 3 cm
* Negative pregnancy test within 48 hours prior to planned index procedure and willing to use reliable birth control for the next 30 days. Reliable birth control is defined as a chemical or barrier method, including an oral contraceptive, injectable contraceptive, or the combination of a spermicide and condoms

Exclusion Criteria:

* Known or suspected cancer, including breast, endometrial, and ovarian
* Subject has Type 2 myoma
* Contraindication and/or allergy to local anesthetic, or oral medications specified in the treatment protocol
* Subject has a history of chronic narcotic use
* Previous uterine artery embolization or other uterine artery occlusion procedure (Doppler or laparoscopic)
* Subject with blood borne pathogens-HIV, hepatitis B, CJD, etc.
* Subject plans to become pregnant within the study period
* Subject has an IUD at the time of the procedure. A subject may be enrolled in the study if the IUD is removed prior to the treatment procedure
* Subject is taking an anticoagulant or antiplatelet medication other than low dose aspirin
* Active pelvic inflammatory disease or pelvic/vaginal infection
* Subject has a known or suspected coagulopathy or bleeding disorder
* Subject has a history of unmanaged endocrine disease
* Subject has current or past, acute or chronic psychiatric disorder which, in the opinion of the Investigator, may preclude proper evaluation and follow-up
* Subject has history of auto-immune, inflammatory, or connective tissue disease
* Subject has a history of disease which increases the risk for fluid overload (i.e. significant cardiac, hepatic, or renal dysfunction)
* Uncontrolled hypertension lasting two years or more
* Use of any experimental drug or device within 30 days prior to the screening visit
* The subject has a terminal illness that may prevent the completion of any follow-up assessments
* Any employee or relative of an employee of the Sponsor company or any Investigator site employee or relative of employees working on the study
* Subject has other co-morbid condition(s) that, in the opinion of the Investigator, could limit the subject's ability to participate in the study or impact the scientific integrity of the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Subject tolerance of procedure-related pain rated on an 11 point scale (0-10) | Immediately post treatment

SECONDARY OUTCOMES:
Subject assessment of most severe post-procedural pain rated on an 11 point scale | Prior to subject discharge from office/day surgery unit
Subject assessment of most severe pain experienced during 48 hours post procedure, rated on an 11 point scale | 48 hours (+ 24 hours) post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Lukes, MD, Principal Investigator — Carolina Women's Research and Wellness Center
Locations (5):
- United States (5):
  - Phoenix Gynecology Consultants, Phoenix, Arizona
  - Florida Woman Care, Boca Raton, Florida
  - Wayne State University, Detroit, Michigan
  - Minnesota Gynecology and Surgery, Edina, Minnesota
  - Carolina Women's Research and Wellness Center, Durham, North Carolina